CLINICAL TRIAL: NCT07164339
Title: Association Between Intraoperative Perfusion Index and Mortality
Brief Title: Intraoperative Perfusion Index and Mortality
Status: Active, not recruiting | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Frederik Lau, MD, Copenhagen University Hospital, Hvidovre
Other Study IDs: F-24084045
Record Dates: First submitted 2025-08-25; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hemodynamic; Perfusion Index; Intraoperative Hemodyamic Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will use routinely collected perioperative data to examine the relationship between intraoperative perfusion index and postoperative outcomes, including mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age who underwent general anesthesia for non-cardiac surgery of any type

Exclusion Criteria:

* No registration of intraoperative perfusion index or no information on vital status 30 days after surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We include every adult patient who underwent general anesthesia for non-cardiac surgery of any type in Danish hospitals in The Capital and Zealand Regions from January 2017 - December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 425000 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days from time of surgery

SECONDARY OUTCOMES:
Composite Adverse Outcome | 30 days from time of surgery
  Proportion of participants who experience ≥1 of the following within 30 days after index surgery:
  1. Postoperative admission to the intensive care unit
  2. Reoperation (within 30 days)
  3. Prolonged length of stay, defined as length of stay falling within the highest (75th-100th) percentile for the patient's surgical category
  4. Acute kidney injury according to Kidney Disease: Improving Global Outcome (KDIGO) criteria (≥1.5-fold increase from baseline within 7 days after surgery or 0.3 mg dl-1 increase within 48 h)
Postoperative ICU Admission | 30 days from date of surgery
  Any ICU admission occurring after index surgery and within 30 days.
Reoperation | 30 days from date of surgery
  Any return to the operating room within 30 days of index surgery.
Prolonged Length of Stay (LOS) | Through hospital discharge (max. 6 months from surgery date)
  Proportion of participants whose index-hospitalization LOS (days from surgery to discharge) falls in the 75th-100th percentile for their surgical category, determined from the study cohort distribution and assessed at discharge.
Acute Kidney Injury | 30 days from date of surgery
  AKI defined by KDIGO criteria (≥1.5× baseline serum creatinine within 7 days or ≥0.3 mg/dL increase within 48 h) occurring within 30 days of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai B Foss, Prof, Study Director — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital - Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No
Data cannot be made available due to ethical and regulatory restrictions.

REFERENCES:
- [Background] Krone S, Bokoch MP, Kothari R, Fong N, Tallarico RT, Sturgess-DaPrato J, Pirracchio R, Zarbock A, Legrand M. Association between peripheral perfusion index and postoperative acute kidney injury in major noncardiac surgery patients receiving continuous vasopressors: a post hoc exploratory analysis of the VEGA-1 trial. Br J Anaesth. 2024 Apr;132(4):685-694. doi: 10.1016/j.bja.2023.11.054. Epub 2024 Jan 19. PMID 38242802
- [Background] Agerskov M, Thusholdt ANW, Holm-Sorensen H, Wiberg S, Meyhoff CS, Hojlund J, Secher NH, Foss NB. Association of the intraoperative peripheral perfusion index with postoperative morbidity and mortality in acute surgical patients: a retrospective observational multicentre cohort study. Br J Anaesth. 2021 Sep;127(3):396-404. doi: 10.1016/j.bja.2021.06.004. Epub 2021 Jul 3. PMID 34226038

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-08-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT07164339/SAP_000.pdf